CLINICAL TRIAL: NCT03969355
Title: Mortality in Tertiary Paediatric Critical Care Centre 2008-2012 Versus 2013-2017: Retrospective Cohort Trial
Brief Title: Mortality in Paediatric Intensive Care
Acronym: Paedmort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, assoc.prof.MD,Ph.D, Brno University Hospital
Other Study IDs: KDAR FN Brno 2019/4
Record Dates: First submitted 2019-05-25; First posted 2019-05-31 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Morbidity, Multiple
Keywords: Paediatric; Intensive care; Mortality
MeSH Terms: interventions — Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paediatric patients 2008-2012: Paediatric patients admitted to intensive care in 2008-2012 who died during PICU stay
  Interventions: Other: Mortality
- Paediatric patients 2013-2017: Paediatric patients admitted to intensive care in 2013-2017 who died during PICU stay
  Interventions: Other: Mortality

INTERVENTIONS:
Other: Mortality — Patients who died during PICU stay

SUMMARY:
Mortality of paediatric patients in intensive care can be considered as on of the parameters of quality of care. Together with the advance in research and medicine there should be a trend towards mortality reduction, however actual data in Czech Republic are not well documented. The aim of this retrospective cohort trial was to evaluate the mortality of paediatric intensive care patients admitted to Department of paediatric anaesthesiology and intensive care between two periods 2008-2012 and 2013 and 2017

DETAILED DESCRIPTION:
Mortality of paediatric patients in intensive care can be considered as on of the parameters of quality of care. Together with the advance in research and medicine there should be a trend towards mortality reduction, however actual data in Czech Republic are not well documented. The aim of this retrospective cohort trial was to evaluate the mortality of paediatric intensive care patients admitted to Department of paediatric anaesthesiology and intensive care between two periods 2008-2012 and 2013 and 2017. The patients records was retrospectively searched and the mortality was adjusted according to the primary admission diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients admitted to intensive care in selected time period

Exclusion Criteria:

* Insufficient documentation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Paediatric patients admitted to the intensive care in selected period (2008-2012. versus 2013-2017).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-05-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Paediatric intesive care unit mortality | During Paediatric intesive care unit (PICU) stay Paediatric patients admitted to the intensive care in selected period (2008-2012. versus 2013-2017)
  Mortality of paediatric patients in selected period in intensive care

SECONDARY OUTCOMES:
Paediatric intesive care unit adjusted mortality | During Paediatric intesive care unit (PICU) stay Paediatric patients admitted to the intensive care in selected period (2008-2012. versus 2013-2017)
  Mortality of paediatric patients in selected period in intensive care according to the admission diagnose and severity of disease

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, assoc.Prof.MD.Ph.D, Study Chair — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided